CLINICAL TRIAL: NCT00397735
Title: Effect of N-acetylcysteine in Preventing Adverse Neonatal Outcomes in Women With Intra-amniotic Infection/Inflammation
Brief Title: N-acetylcysteine in Intra-amniotic Infection/Inflammation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Catalin S Buhimschi, MD, Professor of Obsterics and Gynecology; Frederick Zuspan Endowed Chair, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0603001228
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Labor, Premature; Preterm Premature Rupture of the Membranes; Infection; Inflammation; Chorioamnionitis
Keywords: pregnancy; chorioamnionitis; preterm labor; preterm premature rupture of the membranes; Intra-amniotic infection; Intra-amniotic inflammation
MeSH Terms: conditions — Obstetric Labor, Premature; Preterm Premature Rupture of the Membranes; Infections; Inflammation; Chorioamnionitis | interventions — Amniocentesis; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetylcysteine (Experimental): The subjects enrolled in our research protocol must have evidence of infection/inflammation at amniocentesis in order to receive N-acetylcysteine. Women with positive amniocentesis results The dose of N-acetylcysteine is the one recommended to be used in humans to prevent acetaminophen toxicity: 150 mg/kg loading dose (60 min), followed by 50mg/kg IV continuous infusion rate for 4 hours, and followed by 100 mg/kg IV continuous infusion rate for the following 16 hours. Acetadote (Cumberland Pharmaceuticals) is the only FDA-approved intravenous N-acetylcysteine formulation and will be used in our study.
  Interventions: Procedure: amniocentesis; Drug: N-acetylcysteine or placebo
- Placebo (Placebo Comparator): The subjects enrolled in our research protocol must have infection/inflammation in order to be randomized to receive N-acetylcysteine or placebo. Placebo-assigned patients will receive sodium chloride solution without N-acetylcysteine
  Interventions: Procedure: amniocentesis; Drug: N-acetylcysteine or placebo

INTERVENTIONS:
Procedure: amniocentesis — Amniotic fluid will be retrieved for routine amniocentesis to rule-out or confirm intra-amniotic infection and /or inflammation. The amniocentesis procedure will be clinically indicated and the patient will undergo the procedure independent of our study.
  Other Names: transabdominal amniocentesis
Drug: N-acetylcysteine or placebo — Only women with amniocentesis results consistent with infection/inflammation will be randomized
  Other Names: Mucomyst; Acetadote

SUMMARY:
The aim of the study is to determine if N-acetylcysteine (a potent free radical scavenger) prevents the occurrence of adverse neonatal outcomes in preterm deliveries complicated by infection associated with preterm labor or preterm premature rupture of membranes (PPROM). The working hypothesis is that in pregnancies complicated by intra-amniotic infection or inflammation, N-acetylcysteine protects the fetus by preventing the development, or decreasing the intensity and/or progression of the fetal inflammatory syndrome.

DETAILED DESCRIPTION:
Despite extensive research, the etiology of most preterm births remains unknown. There are significant fetal consequences associated with preterm birth, which include necrotizing enterocolitis, fetal respiratory distress and intra-ventricular hemorrhage. Perinatal mortality is about 44%, 11% and 5% when deliveries occur between 25-28 weeks, 29-32 weeks and 33-34 weeks, respectively. While for many years, it was assumed that the cause of the high morbidity associated with prematurity was the birth of a neonate with a restricted adaptive capacity, it has also been suggested that part of the high perinatal morbidity was the consequence of adverse processes affecting the fetus in utero, rather than of prematurity per se. Intra-amniotic inflammation present in utero early in gestation may trigger the cascade of events leading to preterm birth (i.e. rupture of membranes, cervical ripening, uterine contractions) and provide an intrauterine milieu which is unfavorable or even harmful to the fetus.

Most living organisms have developed well-integrated, antioxidant defenses to scavenge free radicals and control their intracellular concentration. A loss of balance between free radicals and antioxidants (the redox balance) is one mechanism of cell injury in diseases associated with inflammation. N-acetylcysteine is an approved anti-oxidant medication drug used during pregnancy for treatment of mothers with acetaminophen (Tylenol) toxicity. N-acetylcysteine has been safely administered during pregnancy in over 100 women who overdosed with Tylenol and to preterm and healthy term newborns for other purposes. It is a goal of our trial to prevent free radical formation by administering N-acetylcysteine and to further study whether the outcome of preterm deliveries will improve compared to a control group which will not receive placebo infusion

ELIGIBILITY:
Inclusion Criteria:

* Women admitted onto the Labor and Birth Ward or Maternal Special Care Units of the Yale New Haven Hospital who have a clinically indicated amniocentesis which demonstrates presence of intra-amniotic infection and/or inflammation.

Exclusion Criteria:

* Patients that require immediate intervention or close medical supervision (cardiac and renal disease, congestive heart failure, history of asthma), maternal infection (HIV, hepatitis B or C), cord prolapse, known fetal malformation, allergic reactions to N-acetylcysteine, preeclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-10-01; Primary Completion 2012-10-29 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
composite of mortality and severe short term neonatal morbidities (IVH, NEC, BPD, ROP, sepsis, newborn death) | up to 1 year
  IVH, NEC, BPD, ROP, Sepsis, death

SECONDARY OUTCOMES:
neonatal sepsis | up to 30 days
  early and late neonatal sepsis
maternal and umbilical cord plasma antioxidant capacity | up to 1 day
  plasma antioxidant capacity
maternal and umbilical cord plasma N-acetylcysteine levels | up to 1 day
  N-acetylcysteine levels
umbilical cord levels of inflammatory cytokine concentrations | up to 1 day
  pannel of pro and anti inflammatory cytokines
funisitis grades | up to 1 day
  histology
maternal and umbilical cord blood glutathione concentration | up to 1 day
  glutathione levels

CONTACTS AND LOCATIONS:
Overall Officials: Catalin S Buhimschi, MD, MBA, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio